CLINICAL TRIAL: NCT04008589
Title: Non-invasive Current Stimulation for Restoration of Vision (REVIS) After Unilateral Occipital Stroke
Brief Title: Non-invasive Current Stimulation for Restoration of Vision
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Magdeburg (Other)
Collaborators: ERA-NET (Unknown)
Responsible Party: Principal Investigator, Bernhard A. Sabel, Prof., University of Magdeburg
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: REVIS
Record Dates: First submitted 2019-07-03; First posted 2019-07-05 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Stroke; Electrical Stimulation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: randomized, controlled
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- rtACS (Experimental): repetitive transorbital ACS
  Interventions: Device: repetitive transorbital AC Stimulation; Device: combination of transcranial direct current stimulaton and rtACS
- tDCS/rtACS (Experimental): Sequential tDCS - tACS
  Interventions: Device: repetitive transorbital AC Stimulation; Device: combination of transcranial direct current stimulaton and rtACS
- Sham stimulation (Sham Comparator)
  Interventions: Device: repetitive transorbital AC Stimulation; Device: combination of transcranial direct current stimulaton and rtACS

INTERVENTIONS:
Device: repetitive transorbital AC Stimulation — Repetitive transorbital ACS with max 30 Hz, 1,5 mA for 10 days, 20 min/day
Device: combination of transcranial direct current stimulaton and rtACS — Sequential tDCS (anodal occipital stimulation with 2 mA for 20 min/day for 10 days) and rtACS

SUMMARY:
The aim of the study is to evaluate effects of current stimulation of the brain on vision parameters, vision-related quality of life, and physiological parameters to uncover mechanisms of vision restoration. These include EEG-spectra and coherence measures, and visual evoked potentials. The design of stimulation protocols involves an appropriate sham-stimulation condition and sufficient follow-up periods to test whether the effects are stable. This is the first application of non-invasive current stimulation for vision rehabilitation in stroke-related visual field deficits.

ELIGIBILITY:
Inclusion Criteria:

* HH due to ischemic or hemorrhagic stroke
* age between 18 and 75 years
* lesion age at least 6 months
* stable visual field defect across baseline measurement (subjects with spontaneous fluctuations and recovery of vision excluded)
* presence of residual vision and detectable gradual transition between the intact and the absolutely blind part of the visual field according to evaluation of the clinician
* best corrected visual acuity at least 0.4 (20/50 Snellen) or better

Exclusion Criteria:

* known active malignancy
* eye or central nervous system diseases that interfere with the study (including poorly controlled glaucoma)
* electric or electronic implants (e.g. heart pacemaker)
* metal artifacts in the eyes or head (with the exception of dental prosthesis or shunts)
* expected low compliance (e.g. in case of known psychiatric disease, known drug abuse, and dementing syndromes)
* epileptic seizure within the last 10 years
* use of antiepileptic or sedative drugs

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2016-03-31 (Actual); Study Completion 2020-11-05 (Actual)

PRIMARY OUTCOMES:
Size of the visual field | 2 weeks
  Mean threshold in standard static perimetry and and detection accuracy in HRP

SECONDARY OUTCOMES:
Resting EEG power spectra | 2 weeks
  EEG measurement using 128 channel

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Medical Psychology, Magdeburg, Germany

IPD SHARING:
Plan to Share IPD: Yes
Research data will be avalaible without restriction
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After the publication of the data
Access Criteria: Contact to the PI